CLINICAL TRIAL: NCT06603285
Title: A Multi-center, Prospective Study to Observe the Safety, Tolerability, and Efficacy of Remodulin® in Patients With Pulmonary Arterial Hypertension
Brief Title: A Study to Observe the Safety, Tolerability, and Efficacy of Remodulin
Status: Not yet recruiting | Type: Observational
Sponsor: Excelsior (Industry)
Responsible Party: Sponsor
Other Study IDs: EB057-PMS-01
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Treprostinil — sc/iv continuously
  Other Names: Remodulin

SUMMARY:
This is a multi-center, single-arm, prospective study to enroll patients diagnosed as pulmonary arterial hypertension. The objective in this study is to observe the efficacy and safety of treprostinil in subjects with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective study to enroll patients diagnosed as pulmonary arterial hypertension. The expected study period will be 2 years. PAH patients, who met NHI criteria, to receive treprostinil subcutaneously/ intravenously, will be invited to join this study for observation. The dosage and administration schedule of study medication will be judged by investigators. If the eligibility criteria have been met and the subject have signed the informed consent, the subjects will be enrolled into this study. There will be 10 visits: Visit 1 (Screening visit, Week -2 ~ -1), Visit 2 (Week 1, initial of use treprostinil), Visit 3 to 9 (Week 13 to 85), Visit 10 (Week 97). The Day 1 in Week 1 should be the start day of treprostinil treatment. Subjects will be returned to the clinics every 3 months (i.e. 12 weeks) after Visit 2. The NT-proBNP level, WHO functional class, 6-minute walk distance, echocardiography, pulse oximetry, modified Borg Dyspnea Scale, SF-36 questionnaire, and dosage regimens of treprostinil (including dose adjustment) will be collected. For time to clinical worsening and death, it will be followed up during study period. All intercurrent events within 24 months will be recorded. Safety information, including vital signs, and physical exams will be checked. Adverse events of special interest (AESIs) will be reviewed every visit by using a predesignated AESI checklist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic idiopathic or heritable PAH classified as WHO functional class III and IV symptoms.
* PAH patient, who met NHI criteria, will be scheduled to receive subcutaneous/intravenous treprostinil treatment.
* Ability to adhere to the study visit schedule and understand and comply with all protocol requirements.
* Will provide completed and signed written informed consents

Exclusion Criteria:

* Active treatment with injectable prostanoids different from subcutaneous/intravenous treprostinil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who were diagnosed with symptomatic idiopathic or heritable PAH classified as WHO functional class III and IV symptoms and met NHI criteria, will be scheduled to receive subcutaneous/intravenous treprostinil treatment
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NT-proBNP | Week 97
  Calculate the "N terminal pro B type natriuretic peptide" change from baseline to Week 97
Change from baseline in WHO functional class | Week 97
  Calculate the World Health Organization functional class change from baseline to Week 97.
  The World Health Organization (WHO) functional class describes how severe a patient's pulmonary hypertension (PH) symptoms are.
  There are four different classes - I is the mildest and IV is the most severe form of PH.

SECONDARY OUTCOMES:
Time to clinical worsening and death | 96 weeks
  Record the time to clinical worsening and death
Change from baseline in NT-proBNP | Week 13, 25, 37, 49, 61, 73, and 85
  Calculate the change from baseline in NT-proBNP at Week 13, 25, 37, 49, 61, 73, and 85
Change from baseline in 6-minute walk distance (6MWD) | Week 25, 49, 73, and 97
  Calculate the cange from baseline in 6-minute walk distance (6MWD) at Week 25, 49, 73, and 97
Trend of dose usage from initiation treatment to clinical worsening | 96 weeks
  Record all the daily doses which the patients administered during the whole study period
Adverse events of special interest (AESIs) | 96 weeks
  AESIs include infusion site pain, infusion site reaction, headache, diarrhea, nausea, rash, jaw pain, hot flashes, vasodilation, and edema
Change from baseline in WHO functional class | Week 13, 25, 37, 49, 61, 73, and 85
  Calculate the change from baseline in WHO functional class at Week 13, 25, 37, 49, 61, 73, and 85 The World Health Organization (WHO) functional class describes how severe a patient&amp;#39;s pulmonary hypertension (PH) symptoms are.
  There are four different classes - I is the mildest and IV is the most severe form of PH.
Change from baseline in right atrium (RA) area | Week 25, 49, 73, and 97
  RV structure and function will be monitored by echocardiography, including Right atrium (RA) area.
Change from baseline in TAPSE/sPAP ratio. | Week 25, 49, 73, and 97
  RV structure and function will be monitored by echocardiography, including Tricuspid annular plane systolic excursion (TAPSE) / systolic pulmonary artery pressure (sPAP) ratio.
Change from baseline in Pericardial effusion. | Week 25, 49, 73, and 97
  RV structure and function will be monitored by echocardiography, including Pericardial effusion.
Change from baseline in modified Borg Dyspnea Scale | Week 25, 49, 73, and 97
  Calculate the change from baseline in modified Borg Dyspnea Scale at Week 25, 49, 73, and 97.
  The modified Borg Dyspnea scales are patient self-reported measures of one's difficulty in breathing upon exertion. The Scale is a categorical scale with a score from 0 to 10, where 0 represents normal breathing and 10 represents maximum dyspnea.
Change from baseline in SF-36 questionnaire | Week 25, 49, 73, and 97
  Calculate the change from baseline in SF-36 questionnaire at Week 25, 49, 73, and 97.
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.
  It comprises 36 questions that cover eight domains of health. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL.
Intercurrent event | 96 weeks
  Intercurrent events includes consent withdrawn, use of rescue medication, discontinuation from treprostinil treatment, PAH unrelated hospitalization, switch to other PAH drugs (other than treprostinil), add-on PAH drugs, or new-onset co-morbidity.

IPD SHARING:
Plan to Share IPD: No